CLINICAL TRIAL: NCT02073123
Title: A Phase 1/2 Study of the Concomitant Administration of Indoximod Plus Immune Checkpoint Inhibitors for Adult Patients With Advanced or Metastatic Melanoma
Brief Title: Study of IDO Inhibitor in Combination With Checkpoint Inhibitors for Adult Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NLG2103
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Metastatic Melanoma; Stage III Melanoma; Stage IV Melanoma
Keywords: Metastatic melanoma; Stage III melanoma; Stage IV melanoma; unresectable
MeSH Terms: conditions — Melanoma | interventions — 1-methyltryptophan; Ipilimumab; Nivolumab; pembrolizumab

ARMS (3):
- Indoximod + Ipilimumab (Experimental): Indoximod will be administered at 1200mg BID by mouth.
  Ipilimumab administered intravenously at 3 mg/kg every three weeks for a total of four doses.
  Indoximod and ipilimumab will be dosed concurrently. Indoximod will be dosed twice daily on all days of each 21 day cycles (segment 1). Ipilimumab will be dosed on the 1st day of each 21 day cycle for the first 4 cycles. Indoximod dosing will continue after all 4 doses of ipilimumab are administered (segment 2, 28-day cycles).
  Patients will continue until they experience disease progression or limiting toxicity.
  Interventions: Drug: Indoximod; Drug: Ipilimumab
- Indoximod + Pembrolizumab (Experimental): Indoximod will be administered at 1200mg BID by mouth.
  Pembrolizumab administered intravenously at 2 mg/kg every three weeks.
  Interventions: Drug: Indoximod; Drug: Pembrolizumab
- Indoximod + Nivolumab (Experimental): Indoximod will be administered at 1200mg BID by mouth.
  Nivolumab administered intravenously at 240 mg every 2 weeks.
  Interventions: Drug: Indoximod; Drug: Nivolumab

INTERVENTIONS:
Drug: Indoximod — Initial dose of 600mg BID by mouth with escalation planned to 1200mg BID by mouth
  Dose escalation:
  * If 0 of the 3 subjects forming the first cohort experience RLT, 1200mg BID cohort will be enrolled
  * If 1 of the 3 subjects in any cohort experiences a RLT, then enrollment into that cohort will increase to a total of 6 subjects
  * If > 1 of the 3-6 subjects experience a RLT, then the MTD has been exceeded and further enrollment into the cohort will cease
  * If >1 subject at 600mg BID experiences a RLT, the dose will be de-escalated to 400mg BID. If >1 subject at this level experiences a RLT, one additional de-escalation to 200mg BID is allowed
  Dosing cycles are 21 days in length during the combination immunotherapy component (first 4 cycles) and 28 days during indoximod monotherapy. Patients will continue until they experience disease progression or limiting toxicity
  Phase 2 Treatment Plan (Cohort 2) Will receive fixed dose of indoximod determined in phase 1
  Other Names: 1-methyl-D-tryptophan; D-1MT
Drug: Ipilimumab — Ipilimumab administered intravenously at 3 mg/kg every three weeks for a total of four doses.
  Other Names: YERVOY; MDX-010; MDX-101
  Arms: Indoximod + Ipilimumab
Drug: Nivolumab — Nivolumab administered intravenously at 240 mg every 2 weeks.
  Arms: Indoximod + Nivolumab
Drug: Pembrolizumab — Pembrolizumab administered intravenously at 2 mg/kg every three weeks.
  Arms: Indoximod + Pembrolizumab

SUMMARY:
To evaluate the preliminary efficacy of the established dose of indoximod in combination with immune checkpoint inhibition as measured by the best overall response rate (ORR) (complete response (CR) + partial response (PR))across both standard of care agents administered sequentially in patients with unresectable stage III or stage IV melanoma

DETAILED DESCRIPTION:
The incidence of melanoma is increasing. Based upon data obtained between 2004 and 2006, the lifetime probability of developing melanoma in the United States is estimated to be 1 in 37 for men and 1 in 56 for women. In the United States, melanoma is the fifth leading cancer in men and the seventh in women. Locally confined, fully-resectable disease may be curable with current therapy; but Stage IV metastatic disease (or relapsed/recurrent disease) is highly refractory to therapy. Thus, experimental clinical trials provide an accepted treatment option for metastatic or relapsed/refractory melanoma.

The current study is designed as a prospective trial to evaluate the combination of indoximod and checkpoint inhibitors in adult patients with metastatic melanoma. Ipilimumab, pembrolizumab and nivolumab will be used at the recommended approved doses for this indication.

The current trial will be done in two phases: a Phase 1b dose escalation of indoximod in combination with ipilimumab, starting at half the recommended single-agent dose, to establish the recommended Phase 2 dose for the combination.

This will be followed by a three arm expansion study testing a fixed dose of indoximod (at the recommended Phase 2 dose) combined with standard-dose ipilimumab, pembrolizumab or nivolumab.

Treatment will be administered on an outpatient basis. No investigational or commercial cancer directed agents or therapies other than those described below may be administered.

Safety assessment will follow the guidelines provided in the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version.4.03.

Patients will be followed both clinically and radiographically starting 12 weeks after initiation of treatment then every 8 weeks for tumor evaluation. Post-treatment scans will be compared to the baseline scan and responses will be assessed based using mWHO and immune related response criteria (irRC) described by Wolchok et al. (Wolchok et al., 2009).

ELIGIBILITY:
Inclusion Criteria:

* Unresectable Stage III or Stage IV melanoma.
* Patients must have measurable disease, defined as lesions that can be accurately measure in in 2 perpendicular diameters with at least one diameter > 20mm and the other >10mm on conventional CT or MRI or 10mm x 10 mm by spiral CT.
* No systemic treatment in the previous 28 days.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of ipilimumab or indoximod in patients <18 years of age, children are excluded from this study.
* ECOG performance status ≤2 (Karnofsky ≥60% )
* Patients with known brain metastases will only be eligible after their tumors have been treated with definitive resection and/or radiotherapy and they are neurologically stable for at least 1 month off steroids.

Exclusion Criteria:

* Patients who have had molecular targeted therapy (including vemurafenib) or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients who have had prior therapy with immune checkpoint inhibition or or indoximod are excluded from the trial.
* Any other cancer, unless the patient has been disease-free for ≥5 years
* Patients with laboratory evidence of pancreatitis are excluded.
* Patients with autoimmune disease
* Chronic use of immune-suppressive drugs (ie, systemic corticosteroids used in the management of cancer or non-cancer related illnesses, eg, COPD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Overall Incidence of Adverse Events as a Measure of Safety and Tolerability | 17 months
  Phase 1 component:
  Evaluate the safety (adverse events - type, incidence, severity, duration, causality and treatment intervention) of the combination of indoximod and ipilimumab when given concomitantly.
  The safety and tolerability ipilimumab followed by Indoximod will be assessed by listing the overall incidence of AEs. The AEs will be summarized and classified by body system and by treatment group. The type, incidence, severity, and causality of each AE, the duration of the event, and any required treatment interventions will be tabulated. Physical examination results will be presented in the patient data listings. The DLT will be listed per dose level and treatment along with overall frequencies. The data from the expansion part (Phase II) will be used for this part of safety and tolerability assessment.
Phase 2 Dosing | 22 months
  Phase 1 component:
  To determine the recommended Phase 2 dose of indoximod in combination with ipilimumab in patients with unresectable melanoma.
  A minimum of nine patients will be treated depending on DLT. Each dose will be administered to a cohort of 3 patients. If 0 out of 3 or less than 2 out of 6 patients experienced a DLT at any given dose level, the dose escalation will proceed to the next dose level. The MTD is generally the largest dose level at which at most 1 out of 6 patients experiences a DLT. IF DLT is not reached at the highest dose level (1200mg twice daily), no further escalation will proceed and this dose level will be declared the recommended Phase II dose
Overall Response Rate | 22 months
  Phase 2 component:
  To evaluate the preliminary efficacy of the established dose of indoximod in combination with immune checkpoint inhibition as measured by the best overall response rate in patients with unresectable Stage III or Stage IV melanoma.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 22 months
  Adverse event profile of ipilimumab and indoximod in patients with unresectable stage III or Stage IV melanoma participating in phase II portion of the study will be listed, summarized classified by body system. The type, incidence, severity, and causality of each AE, the duration of the event, and any required treatment interventions will be tabulated. Physical examination results will be presented in the patient data listings. The data from the expansion part (Phase II) will be used for this part of safety and tolerability assessment
Overall Survival | 24 months
  b) To evaluate the overall survival (OS) of patients with unresectable stage III or Stage IV melanoma receiving ipilimumab and indoximod. OS, defined as the time between the first dose of study therapy and death (subjects who have not died will be censored at the most recent last-known-alive date), will also be analyzed. The OS rate along with its 95% confidence interval will be presented.
Mechanisms of activity/resistance to IDO/CTLA-4 inhibitor therapy | 24 months
  The mechanisms of activity/resistance to IDO/CTLA-4 inhibitor therapy will be demonstrated through correlative studies.
Progression Free Survival | 22 months
Disease control rate | 22 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Augusta University, Augusta, Georgia
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - New Mexico Cancer Center Alliance, Albuquerque, New Mexico
  - Penn State Hershey Cancer Institue, Hershey, Pennsylvania
  - Huntsman Cancer Institute, Salt Lake City, Utah